CLINICAL TRIAL: NCT06291415
Title: A Multicenter, Phase 1b Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of HMPL-523, a Syk Inhibitor, in Adult Subjects With Immune Thrombocytopenia
Brief Title: The Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of HMPL-523 in Adult Subjects With Immune Thrombocytopenia (ITP)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-523-GLOB1
Record Dates: First submitted 2024-02-13; First posted 2024-03-04 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Immune Thrombocytopenia; Blood Platelet Disorder; Hematologic Diseases; Purpura, Thrombocytopenic; Purpura; Blood Coagulation Disorder; Thrombotic Microangiopathies; Hemorrhagic Disorders; Autoimmune Diseases; Immune System Diseases; Hemorrhage; Pathologic Processes; Skin Manifestations; Thrombocytopenia; Purpura, Thrombocytopenic, Idiopathic; Primary Immune Thrombocytopenia; ITP - Immune Thrombocytopenia
Keywords: ITP; sovleplenib
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Blood Platelet Disorders; Hematologic Diseases; Purpura, Thrombocytopenic; Purpura; Blood Coagulation Disorders; Thrombotic Microangiopathies; Hemorrhagic Disorders; Autoimmune Diseases; Immune System Diseases; Hemorrhage; Pathologic Processes; Skin Manifestations; Thrombocytopenia

STUDY DESIGN:
Intervention Model Description: Part 1: Dose escalation stage - subjects will receive one of 3 dose levels of HMPL-523 to determine the recommended dose of HMPL-523 for the randomized dose optimization- stage (Part 2)
  Part 2: subjects will be randomized in a 1:1 ratio between the 2 dose levels recommended by the SRC to better understand the exposure/efficacy/toxicity relationship. At the end of Part 2, the SRC will evaluate the safety, tolerability, preliminary efficacy, and PK data to determine the Recommended Phase 3 dose (RP3D) of HMPL-523.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): Part 1 will consist of the following 3 dose levels: 300, 400, and 500 mg once daily (QD).
  Interventions: Drug: HMPL-523
- Dose optimization stage (Experimental): In part 2 subjects will be randomized in a 1:1 ratio between the 2 dose levels selected at the end of part 1.
  Interventions: Drug: HMPL-523

INTERVENTIONS:
Drug: HMPL-523 — Syk inhibitor
  Other Names: sovleplenib

SUMMARY:
This is an open-label, multicenter study to evaluate the safety, tolerability, and efficacy of HMPL-523 in adult subjects with ITP.

DETAILED DESCRIPTION:
This study is a Phase 1b, open-label, multicenter, single-arm study to evaluate the safety, tolerability, and preliminary efficacy of HMPL-523 in adult subjects with primary ITP diagnosed at least 3 months prior to enrollment or randomization.

In the dose escalation stage (Part 1), subjects will receive one of 3 dose levels of HMPL-523 to determine the recommended dose of HMPL-523 for the randomized dose optimization- stage (Part 2).

At the end of Part 1, 2 dose levels will be selected to be used in the dose-optimization stage (Part 2) of the study. In Part 2 of the study, subjects will be randomized in a 1:1 ratio between the 2 dose levels to better understand the exposure/efficacy/toxicity relationship.

At the end of Part 2, the Recommended Phase 3 dose (RP3D) of HMPL-523 will be determined based on the safety, efficacy and PK data.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be enrolled in this study only if they satisfy all the following criteria:

1. Adult male or female subjects ≥18 years of age
2. Diagnosis of ITP, with a duration of disease of at least 3 months prior to randomization or enrollment
3. Intolerance or insufficient response or recurrence after at least 1 prior ITP treatment (excluding splenectomy)
4. Response (defined as achieved a platelet count ≥50 × 109/L) to at least 1 prior ITP therapy (including splenectomy)
5. Adequate hematologic, hepatic and renal function

Exclusion Criteria:

Subjects are not eligible for enrollment into this study if any one of the following criteria are met:

1. Evidence of the presence of secondary causes of ITP
2. Clinically serious hemorrhage requiring immediate adjustment of platelets
3. Known history of vital organ transplantation or hematopoietic stem-cell transplantation or chimeric antigen receptor T-cells (CAR-T) therapy
4. Splenectomy within 12 weeks prior to enrollment
5. Presence of active malignancy unless deemed cured by adequate treatment.
6. History of serious cardiovascular disease corrected QT interval (QTcF) ≥450 ms
7. Uncontrolled hypertension
8. Being unsuitable to participate in this study as considered by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of HMPL-523 in adult subjects with primary ITP | week 1 - week 24
  Calculated as the number and percent incidence of participants experiencing adverse events (AE).
Dose Limiting Toxicities | week 1 - week 4
  Defined as an adverse event AE that meets protocol defined Dose Limiting Toxicities (DLT) criteria during the DLT assessment window (first 28 days), unless clearly unrelated to ITP drugs.

SECONDARY OUTCOMES:
Cmax (maximum plasma drug concentration) | week 1 and week 3
  Blood samples will be obtained from all patients to determine maximum plasma drug concentration of HMPL-523 and metabolite M
AUCtau (area under the concentration-time curve over a dosage interval) | week 1 and week 3
  Blood samples will be obtained from all patients to determine area under the concentration time curve over periodic dosing intervals for HMPL-523 and metabolite M1
Tmax (time to reach maximum plasma drug concentration) | week 1 and week 3
  Blood samples will be obtained from all patients to determine time to reach maximum plasma concentration of HMPL-523 and metabolite M1
Cmin (minimum plasma drug concentration) | week 1 - week 20
  Blood samples will be obtained from all patients to determine minimum plasma concentration of HMPL-523 and metabolite M1

CONTACTS AND LOCATIONS:
Overall Officials: William Schelman, MD, PhD, Study Director — Hutchmed
Locations (28):
- United States (10):
  - Childrens Hospital of California, Irvine, California
  - Georgetown University Medical Center - Georgetown Lombardi Comprehensive Cancer Center, Georgetown, Delaware
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - San Juan Oncology Associates, Farmington, New Mexico
  - East Carolina University, Brody School of Medicine, Greenville, North Carolina
  - Taussig Cancer Institute, Cleveland, Ohio
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Texas Oncology San Antonio Medical Center, San Antonio, Texas
  - University of Washington (UW) Medical Center, Seattle, Washington
- Australia (4):
  - Peninsula Private Hospital, Frankston, Victoria
  - The Perth Blood Institute (PBI) Hollywood Specialist Centre, West Perth, Western Australia
  - Royal Adelaide Hospital, Adelaide
  - Canberra Hospital, Canberra
- Germany (4):
  - Charite university, Berlin
  - Marien Hospital Dusseldorf, Düsseldorf
  - UMG Gottingen Hämatologie, Göttingen
  - University Hospital of Schleswig-Holstein, Department of Haematology and Oncology, Lübeck
- Norway (2):
  - Sykehuset Ostfold Kalnes (fosta) / Osfold Hospital Trust (MSL), Grålum
  - Oslo University Hospital, Oslo
- Spain (8):
  - Hospital del Mar Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - University de Burgos, Burgos
  - Hospital Gregorio Maranon Madrid, Madrid
  - Clinica Universidad de Navarra, Madrid
  - Hospital Infanta Leonor, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Morales Meseguer, Murcia